CLINICAL TRIAL: NCT02582879
Title: informCLL™: A Disease Registry for Patients With Chronic Lymphocytic Leukemia
Acronym: informCLL
Status: Completed | Type: Observational
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: PCYC-1134M-CA
Record Dates: First submitted 2015-09-08; First posted 2015-10-21 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Leukemia; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with CLL/SLL: Patients with CLL/SLL in a real-world setting initiating treatment with approved oral kinase inhibitors, BCL-2 inhibitors and other approved anti-CLL therapies/regimens.

SUMMARY:
The study is designed as a multicenter, prospective, observational registry of CLL/SLL patients who are initiating approved oral kinase inhibitors, BCL-2 inhibitors or other approved anti-CLL therapies/regimens. The study will characterize treatment patterns and their association with patient characteristics, healthcare resource utilization, and clinical outcomes, as well as patient-reported outcome (PRO) measures.

DETAILED DESCRIPTION:
This multicenter, prospective, observational registry of CLL patients is designed to characterize and describe treatment patterns for those initiating treatment with approved oral kinase inhibitors and other approved anti-CLL therapies/ regimens. The registry will provide information on regimens used to treat first-line and later lines of CLL as well as the sequencing of treatment regimens. The registry will also evaluate the association of these treatment patterns with patient characteristics, healthcare resource utilization, and functional outcomes including patient-reported HRQoL. These data will provide information to physicians that may help guide clinical practice and appropriate use of therapies, and will also provide information on HRQoL and healthcare resource utilization that will be of interest to healthcare decision makers.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Clinical diagnosis of CLL/SLL that meets published diagnostic criteria (Hallek 2008)
* Initiating anti-CLL/SLL treatment regimen (excluding clinical trials) within ±45 days of enrollment
* Availability of documentation of previous CLL/SLL treatment and duration of response in the patient's medical records if patient has received prior line(s) of treatment (i.e. NOT treatment naïve)
* Willing and able to provide informed consent
* Willing and able to complete PRO instrument
* Willing and able to provide information on patient survey questionnaire
* Willing and able to provide a blood sample at time of enrollment prior to receiving treatment, as possible

Exclusion Criteria:

* Diagnosis of B-cell malignancies other than CLL/SLL
* Estimated life expectancy <6 months
* Currently receiving treatment in an interventional clinical trial at time of entry into this study * Note- Exceptions: 1) Patients may enroll in interventional clinical trials for indications other than CLL/SLL, 2) The interventional clinical trial treatment is not the treatment used for meeting Inclusion Criteria #2 (or "Index Treatment"), 3) Patients may enroll in an interventional clinical trial indicated for CLL/SLL as later line of treatment after discontinuing the Index Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will aim to enroll approximately 1500 patients with CLL/SLL from a total of 200 sites in the US over a 45 month enrollment period. In order to best capture real-world treatment patterns, site recruitment will aim to include approximately 85% of sites from the community hematology-oncology setting.
Sampling Method: Non-Probability Sample
Enrollment: 1504 (Actual)
Dates: Start 2015-09; Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Summarize baseline characteristics of study population, among CLL patients in a real-world setting | up to 7 years
  - Summarize baseline characteristics of study participants
Summarize treatment patterns among CLL patients in a real-world setting | up to 7 years
  * Summarize number of participants on various initial and subsequent treatments
  * Summarize proportion of patients switching therapies at each follow up time point
Summarize clinical outcomes among CLL patients in a real-world setting | up to 7 years
  - Measures of effectiveness used will include survival status, ECOG Health status, response assessments as evaluated by the investigator such as: complete response, partial response, stable disease, progressive disease
Summarize health care resource utilization among CLL patients in a real-world setting | up to 7 years
  - Summarize health care resource utilization among study participants

SECONDARY OUTCOMES:
Summarize non serious adverse events (AEs) that led to discontinuation/modification/interruption of therapy and all serious adverse events in CLL patients | up to 7 years
  - Summarize frequencies and percentages of AEs, that led to discontinuation/modification/interruption of therapy or death in CLL patients
Summarize patient-reported HRQoL scores | up to 7 years
  - Summarize HRQoL scores as measured by FACT-G and additional questions from other PRO instruments at baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alex Young, Study Director — Pharmacyclics LLC.
Locations (190):
- United States (190):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Northwest Alabama Cancer Center, PC, Muscle Shoals, Alabama
  - Arizona Oncology Associates, PC - HAL, Glendale, Arizona
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL-Scottsdale, Tempe, Arizona
  - Mercy Research, Fort Smith, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Clopton Clinic of Jonesboro, Inc., Jonesboro, Arkansas
  - CARTI - Central Arkansas Radiation Therapy Institute, Little Rock, Arkansas
  - John Muir Health, Concord, California
  - North County Oncology Medical Clinic, Oceanside, California
  - Sansum Clinic, Santa Barbara, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Sansum Clinic, Solvang, California
  - Gregory Smith, MD (Private Practice), St. Helena, California
  - Solano Hematology Oncology, Vallejo, California
  - Rocky Mountain Cancer Centers, LLP- Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP- Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP- Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, LLP- Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers, LLP- Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, LLP- Longmont, Longmont, Colorado
  - Rocky Mountain Cancer Centers, LLP- Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers, LLP- Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, LLP- Thornton, Thornton, Colorado
  - University Cancer Institute, LLC, Boynton Beach, Florida
  - Broward Oncology Associates, PA, Fort Lauderdale, Florida
  - Cancer Specialists, LLC, Jacksonville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Lakeland Regional Health Systems Inc, Lakeland, Florida
  - Watson Clinic Cancer and Research Center, Lakeland, Florida
  - Sacred Heart Cancer Center, Pensacola, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Southeast Georgia Physician Associates Hematology & Oncology, Brunswick, Georgia
  - The University of Chicago, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mid-Illinois Hematology & Oncology Associates,Ltd., Normal, Illinois
  - Illinois Cancer Care, P.C., Peoria, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Healthcare Research Network III, LLC, Tinley Park, Illinois
  - St. Vincent Anderson Regional Hospital, Anderson, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Horizon Oncology Research, Inc, Lafayette, Indiana
  - Memorial Medical Group Clinical Research Institute, South Bend, Indiana
  - Good Samaritan Hospital, Vincennes, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Physicians Clinic of Iowa, Cedar Rapids, Iowa
  - Covenant Clinic, Waterloo, Iowa
  - Cotton-O'Neil Clinical Research Center, Hematology and Oncology, Topeka, Kansas
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - West Ky Hematology & Oncology Group, PSC, Paducah, Kentucky
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Christus Cancer Treatment Center, Shreveport, Louisiana
  - Maine Research Associates, Lewiston, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Western Maryland Health System, Cumberland, Maryland
  - Antietam Oncology and Hematology Group PC, Hagerstown, Maryland
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Beth Israel Deaconess Hospital- Plymouth, Plymouth, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - St John Providence Hospital, Novi, Michigan
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - Central Cancer Care Center, Bolivar, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Heartland Regional Medical Center d/b/a Cancer Care St. Joseph Mosaic Life Care, Saint Joseph, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Mary Lanning Healthcare Morrison Cancer Center, Hastings, Nebraska
  - Nebraska Hematology-Oncology, P.C, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Trinitas Hospital, Elizabeth, New Jersey
  - Hematology Oncology Physicians of Englewood, PA, Englewood, New Jersey
  - Meridian Health Systems, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Southern Oncology Hematology Associates, Williamstown, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - St. Francis Hospital, East Hills, New York
  - North Shore Hematology Oncology Associates, PC, East Setauket, New York
  - Hematology Oncology Associates Of Central New York, East Syracuse, New York
  - Glen Falls Hospital Cancer Center, Glens Falls, New York
  - North Shore Long Island Jewish Hospital, Manhasset, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - MHO Research Foundation, Inc., New York, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - White Plains Hospital, White Plains, New York
  - CCS Oncology, Williamsville, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Leo Jenkins Cancer Center/ECU School of Medicine, Greenville, North Carolina
  - Raab Clinic, Morehead City, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Mid Ohio Oncology Hematology, DBA The Mark H. Zangmeister Center, Columbus, Ohio
  - Wright State University, Middletown, Ohio
  - Toledo Community Hospital Oncology Program - CCOP Toledo, Toledo, Ohio
  - St. Elizabeth Hospital, Youngstown, Ohio
  - Mercy Research - Mercy Clinic Oncology and Hematology, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Hematology Oncology Associates, PC, Medford, Oregon
  - Hematology Oncology Associates, Medford, Oregon
  - Compass Oncology- Hoyt, Portland, Oregon
  - Compass Oncology- Barnes, Portland, Oregon
  - Compass Oncology- Broadway, Portland, Oregon
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Compass Oncology- Tualatin, Tualatin, Oregon
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - University Cancer Institute, LLC, Monroeville, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Hematology & Oncology Associates of Northeastern PA, Scranton, Pennsylvania
  - Susquehanna Cancer Center, Williamsport, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Cancer Centers of the Carolinas- Easley, Easley, South Carolina
  - Cancer Centers of the Carolinas- Butternut, Greenville, South Carolina
  - Hematology and Oncology Associates of SC, LLC, Greenville, South Carolina
  - Greenville Hospital System Medical Center, Greenville, South Carolina
  - Greenville Health System, Greer, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas- Spartanburg, Spartanburg, South Carolina
  - Prairie Lakes Hospital, Watertown, South Dakota
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Hendrick Cancer Center, Abilene, Texas
  - Texas Oncology - Abilene, Abilene, Texas
  - Texas Oncology- Allen, Allen, Texas
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncoogy - Arlington North, Arlington, Texas
  - Texas Oncology- Arlington South, Arlington, Texas
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - P.A.- Austin, Austin, Texas
  - South Austin Cancer Center, Austin, Texas
  - Texas Oncology - PA, Beaumont, Texas
  - Texas Oncology, P.A - Beaumont, Beaumont, Texas
  - Texas Oncology-Bedford, Bedford, Texas
  - Texas Oncology - Carrollton, Carrollton, Texas
  - Texas Oncology - Dallas Presbyterian, Dallas, Texas
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - El Paso Cancer Treatment Center- West, El Paso, Texas
  - Texas Oncology - P.A. - El Paso, El Paso, Texas
  - Texas Oncology - El Paso, El Paso, Texas
  - Texas Oncology, P.A.- Flower Mound, Flower Mound, Texas
  - Texas Oncology-Grapevine, Grapevine, Texas
  - Texas Oncology PA, Harlingen, Texas
  - Texas Oncology - P.A.- Longview, Longview, Texas
  - Texas Oncology - P.A.-McAllen, McAllen, Texas
  - Texas Oncology- McKinney, McKinney, Texas
  - Texas Oncology -P.A.- Mesquite, Mesquite, Texas
  - Texas Oncology - P.A.- Midland, Midland, Texas
  - Texas Oncology - P.A.- Odessa, Odessa, Texas
  - Texas Oncology - P.A.- Paris, Paris, Texas
  - Texas Oncology - P.A.- Plano, Plano, Texas
  - Texas Oncology- Plano West, Plano, Texas
  - Texas Oncology - Rockwall, Rockwall, Texas
  - Texas Oncology- San Antonio Downtown, San Antonio, Texas
  - Texas Oncology- San Antonio Northeast, San Antonio, Texas
  - Texas Oncology- San Antonio Stone Oak, San Antonio, Texas
  - Texas Oncology - P.A.-Sherman, Sherman, Texas
  - Texas Oncology - P.A.-Sugar Land, Sugar Land, Texas
  - Tyler Hematology Oncology, Tyler, Texas
  - Texas Oncology-P.A-Tyler, Tyler, Texas
  - Texas Oncology, P.A. - Horizon Circle, Waco, Texas
  - Texas Oncology, P.A. - Waco, Waco, Texas
  - Texas Oncology-P.A.- Webster, Webster, Texas
  - Texas Oncology-Weslaco, Weslaco, Texas
  - Cancer Specialists of Tidewater, Newport News, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
  - Providence Everett Medical Center, Everett, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Multicare Institute for Research and Innovation, Tacoma, Washington
  - Compass oncology, Vancouver, Washington
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - HSHS St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - ProHealth Care, Waukesha, Wisconsin

REFERENCES:
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=PCYC-1134M-CA&Latitude=&Longitude=&LocationName=#additional-resources-section